CLINICAL TRIAL: NCT04358549
Title: Open Label, Randomized, Controlled Phase 2 Proof-of-Concept Study of the Use of Favipiravir Compared to Standard of Care in Hospitalized Subjects With COVID-19
Brief Title: Study of the Use of Favipiravir in Hospitalized Subjects With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAVI-COV-US201
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Standard of Care

STUDY DESIGN:
Intervention Model Description: Open-label, randomized (1:1 ratio) to receive favipiravir plus standard of care or standard of care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Favipiravir Treatment Arm (Experimental): Day 1: favipiravir 1800 mg BID plus Standard of Care (SOC) Days 2-14: 1000 mg BID plus SOC. For subjects with Child-Pugh A liver impairment: Days 2-14: 800 mg BID plus SOC
  Interventions: Drug: Favipiravir
- Standard of Care Arm (Other): Standard of Care for 14 days
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Favipiravir — Favipiravir to be administered as an oral tablet or made into a slurry for subjects who cannot swallow tablets
  Arms: Favipiravir Treatment Arm
Other: Standard of Care — Standard of Care for individual study site as determined by each hospital's protocol
  Arms: Standard of Care Arm

SUMMARY:
To determine the effect of favipiravir + SOC v. SOC on COVID-19 viral clearance.

DETAILED DESCRIPTION:
This is an open label, randomized, controlled, multicenter Phase 2 proof-of-concept study of favipiravir in hospitalized subjects with Corona Virus Disease (COVID) -19. Subjects will be randomized within their study site and stratified by the severity of their disease to receive either favipiravir + standard of care (SOC) or SOC alone.

The dose regimen will be 1800 mg favipiravir bis in die (BID) plus SOC or SOC alone on Day 1 followed by 1000 mg BID favipiravir (800 mg BID for subjects with Child-Pugh A liver impairment) plus SOC or SOC for the next 13 days.

The study will have 14 days of treatment and 46 days of follow-up.

Approximately 50 patients are planned to be enrolled in the trial at approximately 8 study sites in the US.

ELIGIBILITY:
Inclusion Criteria:

1) Adults (18 to 80 years old):

1. within 72 hours of their hospitalization for infection with Severe Acute Respiratory Syndrome - Corona Virus - 2 (SARS-CoV-2), AND,
2. within 72 hours of the latest Polymerase Chain Reaction (PCR) positive result and within 7 days of the 1st PCR positive result for SARS-CoV-2. (The latest PCR could be the only PCR result.), AND,
3. within 10 days of onset of any COVID-19 symptoms.

Exclusion Criteria:

1. Subject has a concomitant bacterial respiratory infection unless cleared by the Sponsor
2. Subject has a history of abnormalities of uric acid metabolism unless cleared by the Sponsor.
3. Subject has a history of hypersensitivity to an anti-viral nucleoside analog drug targeting a viral RNA polymerase
4. Subject is using adrenocorticosteroids (except topical or inhaled preparations or oral preparations equivalent to or less than 10 mg of oral prednisone) or immunosuppressive or immunomodulatory drugs (e.g., immunosuppressants, anticancer drugs, interleukins, interleukin antagonists or interleukin receptor blockers). Dexamethasone 6 mg daily (PO or IV) for 10 days is permitted.
5. Subject has a serious chronic disease (e.g., human immunodeficiency virus (HIV), cancer requiring chemotherapy within the preceding 6 months, moderate or severe hepatic insufficiency and/or unstable renal, cardiac, pulmonary, neurologic, vascular, or endocrinologic disease states requiring medication dose adjustments within the last 30 days).
6. Has previously received favipiravir within the past 30 days
7. Has renal insufficiency requiring hemodialysis or continuous ambulatory peritoneal dialysis (CAPD) or glomerular filtration rate of less than 20 mL/min.
8. Has liver impairment greater than Child-Pugh A.
9. Has a history of alcohol or drug abuse in the previous 6 months.
10. Has a psychiatric disease that is not well controlled where controlled is defined as: stable on a regimen for more than one year.
11. Has taken another investigational drug within the past 30 days.
12. Is on another antiviral or is participating in another clinical trial for the treatment of COVID-19
13. Subject is on a ventilator at the time of study entry
14. Is deemed by the Investigator to be ineligible for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - HonorHealth, Scottsdale, Arizona
  - University of Miami Miller School of Medicine, Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial Health Care, Worcester, Massachusetts
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finberg RW, Ashraf M, Julg B, Ayoade F, Marathe JG, Issa NC, Wang JP, Jaijakul S, Baden LR, Epstein C. US201 Study: A Phase 2, Randomized Proof-of-Concept Trial of Favipiravir for the Treatment of COVID-19. Open Forum Infect Dis. 2021 Dec 7;8(12):ofab563. doi: 10.1093/ofid/ofab563. eCollection 2021 Dec. PMID 34888401

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Favipiravir Treatment Arm | Standard of Care Arm
Started | 25 | 25
ITT Population (Randomized Subjects) | 25 | 25
Safety Population (Patients Who Received Either Favipiravir + SOC or SOC Alone) (One patient randomized in favipiravir + SOC arm withdrew before the first dose of favipiravir.) | 24 | 25
Completed | 15 | 17
Not Completed | 10 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Start remdesivir | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Favipiravir Treatment Arm | Standard of Care Arm | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.37) | 58.9 (13.90) | 57.2 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 17 | 12 | 29
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Smoking Status [Count of Participants; unit: Participants]
  Non-smoker | 17 | 14 | 31
  Ex-smoker | 6 | 11 | 17
  Smoker | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Viral Clearance
Description: To determine the effect of favipiravir + SOC v. SOC on viral clearance of COVID-19 as measured by nasopharyngeal and oropharyngeal sampling
Time Frame: Day 29
Population: ITT
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Favipiravir Treatment Arm | Standard of Care Arm
Number analyzed (Participants) | 25 | 25
days | 16.0 [12.0 to 29.0] | 30.0 [12.0 to 31.0]
Statistical Analysis 1: Comparison: Favipiravir Treatment Arm vs Standard of Care Arm; Test type: Superiority; p = 0.0415, Log Rank; Median Difference (Final Values) = 14

2. Secondary Outcome: Status of Clinical Recovery as Measured by the Study-specific 6-point Ordinal Scale
Description: To determine the clinical benefit of administering favipiravir plus SOC compared to SOC alone, clinical benefit will be measured using a study-specified ordinal scale on Day 15 in adult patients hospitalized with COVID-19.
Time Frame: on Day 15
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir Treatment Arm | Standard of Care Arm
Number analyzed (Participants) | 25 | 25
Participants
  Not Hospitalized | 18 | 18
  Hospitalized, not requiring supplemental oxygen | 1 | 3
  Hospitalized, requiring supplemental oxygen | 4 | 1
  Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0 | 0
  Hospitalized, on invasive mechanical ventilation or ECMO | 1 | 0
  Death | 0 | 0
  Not available | 1 | 3
Statistical Analysis 1: Comparison: Favipiravir Treatment Arm vs Standard of Care Arm; Test type: Superiority; Odds Ratio (OR) = 0.653, 90% CI 2-sided [0.190 to 2.240]

3. Secondary Outcome: Time to the National Early Warning Score 2 (NEWS2) of 2 or Less, or Hospital Discharge
Description: The NEWS2 is based on a simple aggregate scoring system in which a score is allocated to physiological measurements, already recorded in routine practice, when patients present to, or are being monitored in hospital. Six simple physiological parameters form the basis of the scoring system: respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new confusion, temperature. The time to aggregate NEWS2 score of ≤ 2 (sustained for at least 72 hours) or hospital discharge is analyzed.
Time Frame: through Day 29
Population: ITT
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Favipiravir Treatment Arm | Standard of Care Arm
Number analyzed (Participants) | 25 | 25
days | 4.0 [3.0 to 8.0] | 7.0 [4.0 to 10.0]
Statistical Analysis 1: Comparison: Favipiravir Treatment Arm vs Standard of Care Arm; Test type: Superiority; p = 0.9879, Log Rank; Median Difference (Final Values) = 3

4. Secondary Outcome: Characterize the Pharmacokinetics (PK) of Favipiravir in Plasma: Cmax
Description: Measurement of maximum plasma concentration
Time Frame: through Day 14
Population: PK population: All subjects in the safety population that have at least one result that can be used in the PK summaries.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Favipiravir Treatment Arm
Number analyzed (Participants) | 23
µg/mL
  Day 1 | 60.9 [22.0 to 84.5]
  Day 2 | 47.1 [16.7 to 109]
  Day 8: number analyzed (Participants) | 20
  Day 8 | 51.4 [17.1 to 133]
  Day 14: number analyzed (Participants) | 17
  Day 14 | 50.8 [14.2 to 134]

5. Secondary Outcome: Characterized the Pharmacokinetics (PK) of Favipiravir in Plasma: Cmin
Description: Measurement of minimum plasma concentration
Time Frame: through Day 14
Population: PK population: All subjects in the safety population that have at least one result that can be used in the PK summaries.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Favipiravir Treatment Arm
Number analyzed (Participants) | 23
µg/mL
  Day 1 | 3.24 [0.120 to 36.1]
  Day 2 | 8.19 [0.152 to 70.2]
  Day 8: number analyzed (Participants) | 20
  Day 8 | 17.1 [1.04 to 88.4]
  Day 14: number analyzed (Participants) | 17
  Day 14 | 15.5 [0.815 to 87.4]

6. Secondary Outcome: Characterized the Pharmacokinetics (PK) of Favipiravir in Plasma: Area Under Curve (AUC 0-24)
Description: Measurement of the area under the curve of plasma concentration versus time profile
Time Frame: through Day 14
Population: PK population: All subjects in the safety population that have at least one result that can be used in the PK summaries.
Measure: Median (Full Range); unit: hr*µg/mL
Arm/Group | Favipiravir Treatment Arm
Number analyzed (Participants) | 23
hr*µg/mL
  Day 1 | 414 [161 to 1240]
  Day 2 | 488 [135 to 2120]
  Day 8: number analyzed (Participants) | 20
  Day 8 | 786 [189 to 2580]
  Day 14: number analyzed (Participants) | 17
  Day 14 | 772 [151 to 2680]

ADVERSE EVENTS:
Time Frame: Until 60 days from Enrollment
Arm/Group | Favipiravir Treatment Arm | Standard of Care Arm
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/24 | 3/25
Other Adverse Events (participants affected / at risk) | 13/24 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Favipiravir Treatment Arm (N=24) | Standard of Care Arm (N=25)
Osteomyelitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Basal ganglia hemorrhage (Nervous system disorders) | 1 | 0
Necrosis (General disorders) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Favipiravir Treatment Arm (N=24) | Standard of Care Arm (N=25)
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Inflammatory marker increased (Investigations) | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication until earlier of: Sponsor publishes multisite results, Sponsor notice that multisite publication no longer planned, and 18 months after Study close. Submission to Sponsor of proposed publication for 30-45 days prior to submission for publication. Good faith consideration by Site of Sponsor's comments; deletion of any of Sponsor's confidential information. Sponsor may require up to additional 60-day delay to file patent applications for patentable subject matter in the publication.

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT04358549/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT04358549/SAP_001.pdf